CLINICAL TRIAL: NCT06776991
Title: Reward Processing and Exposure Therapy
Brief Title: Reward Processing and Exposure Therapy for Social Anxiety Disorder
Acronym: METER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tomislav Zbozinek, PhD, Assistant Project Scientist, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K23MH133971-01A1 (NIH); 1K23MH133971-01A1 (NIH)
Record Dates: First submitted 2024-11-13; First posted 2025-01-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-01

CONDITIONS: Social Anxiety Disorder (Social Phobia); Public Speaking Anxiety; Anhedonia; ANXIETY DISORDERS (or Anxiety and Phobic Neuroses); Phobic Disorders
Keywords: Exposure Therapy; Anxiety; Social Anxiety; Public Speaking Anxiety; Anhedonia; Reward Processing; Inhibitory Retrieval; Positive Affect Treatment; Relaxation Treatment
MeSH Terms: conditions — Phobia, Social; Anhedonia; Anxiety Disorders; Phobic Disorders | interventions — Implosive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Affect Treatment - Behavioral (PAT-B) (Experimental): Focused on improving reward processing and anhedonia using PAT-B. Expected to reduce negative affect and increase positive affect. Then, exposure therapy to reduce public speaking anxiety.
  Interventions: Behavioral: Positive Affect Treatment - Behavioral (PAT-B); Behavioral: Exposure Therapy
- Relaxation Treatment (Active Comparator): Focused on relaxation and mindfulness using Relaxation Treatment. Expected to reduce negative affect. Then, exposure therapy to reduce public speaking anxiety.
  Interventions: Behavioral: Relaxation Treatment; Behavioral: Exposure Therapy

INTERVENTIONS:
Behavioral: Positive Affect Treatment - Behavioral (PAT-B) — 8 therapy sessions conducted individually with a therapist. Focuses on improving reward processing to increase positive emotional experience. Specific techniques include psychoeducation on mood cycle and positive emotions, mood monitoring, behavioral activation, and imaginal recounting and savoring of behavioral activation events. Intervention includes between-session practice.
  Arms: Positive Affect Treatment - Behavioral (PAT-B)
Behavioral: Relaxation Treatment — 8 therapy sessions conducted individually with a therapist. Focuses on mindfulness and relaxation skills. Specific techniques include mindfulness approaches from dialectical behavior therapy, diaphragmatic breathing, and progressive muscle relaxation. Intervention includes between-session practice.
  Arms: Relaxation Treatment
Behavioral: Exposure Therapy — 8 therapy sessions conducted individually with a therapist using the inhibitory retrieval model of exposure therapy. Sessions are designed to include four exposures each (32 exposures total). Each exposure is a public speech delivered to an audience. Goal of this treatment is to reduce public speaking anxiety. Principles of exposure therapy that will be incorporated are maximizing prediction error, maintaining attention to the situation/stimuli that are perceived predictors of the feared outcome (e.g., social rejection), removing safety signals, variability, engaging in post-exposure rehearsal/consolidation, deepened extinction, and positive occasion setter extinction. Intervention does not include between-session practice.

SUMMARY:
The investigators are conducting a clinical trial of therapy for public speaking anxiety. There are many eligibility criteria, but the main ones are that participants need to be socially anxious and have public speaking anxiety. In this clinical trial, all participants will do exposure therapy. Before doing exposure therapy in the study, though, participants will be randomized to do one of two treatments: i) a positive mood treatment, which is designed to increase how positive people feel, and ii) a relaxation treatment, which is designed to help people feel more relaxed. The investigators are doing this study to see whether doing the positive mood treatment or relaxation treatment first will affect how well exposure therapy works.

DETAILED DESCRIPTION:
A substantial number of individuals do not achieve clinically significant symptom relief from exposure therapy, or they may experience return of fear following completion of exposure therapy. This clinical trial aims to intervene on one potential reason exposure therapy's success is mitigated: anhedonia. Anhedonia is characterized by physiological, behavioral, neural, and self-report deficits in reward processing - where reward processing includes anticipation of reward (positive experiences, such as social connection, food, personal achievement), engaging in effort for reward, feeling motivated for reward, savoring reward when it occurs, taking responsibility for the occurrence of reward, and learning what leads to reward. In basic scientific studies of non-humans and humans, poor reward processing is associated with poor extinction of fear (i.e., poor reduction of fear), and anxiety disorders (e.g., social anxiety disorder) often have elevated anhedonia. Therefore, individuals who are both anxious and anhedonic likely experience deficits in extinguishing fear, which is a core process of exposure therapy. Methods of improving reward processing and anhedonia may thus increase the efficacy of exposure therapy.

The present clinical trial will recruit individuals who are clinically socially anxious, have elevated public speaking anxiety, and have anhedonia / poor reward processing. Participants will all do Exposure Therapy for public speaking anxiety, but before doing so, they will be randomized to one of two treatment conditions: the behavioral portion of Positive Affect Treatment (PAT-B; to increase reward processing and reduce anhedonia), and Relaxation Treatment (comprised of mindfulness, diaphragmatic breathing, and progressive muscle relaxation). Assessments including a public speech behavioral approach task, questionnaires, and fear conditioning. The behavioral approach task and questionnaires will be conducted before participants' first treatment (Pre Tx; before PAT-B or Relaxation Treatment), after their first treatment (Post Tx-1), after Exposure Therapy (Post Tx-2), and three months after completing Exposure Therapy (3-Month Follow-Up). The fear conditioning task will be conducted before participants' first treatment (Pre Tx; before PAT-B or Relaxation Treatment) and after their first treatment (Post Tx-1); this will be done either in an fMRI or non-fMRI setting, depending on whether participant has MRI contraindications or based on study needs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of social anxiety disorder from the Structural Clinical Interview for DSM 5.
* Elevated fear of public speaking, defined as a score of >= 66 (+1SD from the mean of population norms on a scale of 17-85) on the Public Speaking Anxiety Scale (PSAS; Bartholomay, E. M., & Houlihan, D. D. (2016). Public Speaking Anxiety Scale: Preliminary psychometric data and scale validation. Personality and individual differences, 94, 211-215), which is a self-report scale measuring anxiety of public speaking.
* Low reward processing, defined as a score of <56 (less than the population mean) on the Dimensional Anhedonia Rating Scale (DARS) (Rizvi, S. J., Quilty, L. C., Sproule, B. A., Cyriac, A., Bagby, R. M., & Kennedy, S. H. (2015). Dimensional Anhedonia Rating Scale (DARS) [Database record]. APA PsycTests).
* Medication-free or stabilized on psychotropic medications for a minimum standard length of time (1 month for benzodiazepines and beta blockers, 3 months for SRIs/SNRIs and heterocyclics).
* Psychotherapy-free or stabilized on alternative psychotherapies other than cognitive or behavioral therapies that were not focused on their anxiety disorder for at least 6 months prior to study entry.
* Age 18-60.
* Fluent in English.
* To conduct MRI version of fear conditioning task, must have no MRI contraindications.

Exclusion Criteria (none of the following):

* Recent suicidal ideation with intent or plan - defined as suicidal ideation with intent or plan in the past year.
* Lifetime history of suicide attempts.
* History of bipolar disorder, psychosis, intellectual disability, or organic brain damage.
* Substance use disorder within the last 6 months.
* Major respiratory, cardiovascular, pulmonary, neurological, or muscular-skeletal diseases.
* Pregnant or planning to become pregnant for next 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Public Speaking Anxiety Scale (PSAS) | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24). Also Sessions 2, 4, 6, 8 of each therapy (corresponding to ~weeks 1, 2, 3, 4, 7, 8, 9, 10).
  Self-reported public speaking anxiety symptom severity. This measure is a 17-item questionnaire using a 1-5 scale (1 = not at all, 3 = moderately, 5 = extremely) with sum scores ranging 17-83. Higher = worse.
Behavioral Approach Task - Anxiety | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Self-reported anxiety during public speaking Behavioral Approach Task. The Behavioral Approach Task is a task in which the participant gives a speech to a small audience (1-4 people) on a topic of the experimenter's choosing. One of four speech topics will be conducted (counterbalanced). The investigators will measure participants' anxiety throughout this task, including anxiety while anticipating the speech and delivering the speech. Anxiety will be measured "right now" on a 0-100 scale, where 0 = no anxiety, 50 = moderate, and 100 = extreme. Higher = worse.
Behavioral Approach Task - Likelihood Expectancy | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Self-reported likelihood that participant will be / was negatively socially evaluated during public speaking Behavioral Approach Task. The Behavioral Approach Task is a task in which the participant gives a speech to a small audience (1-4 people) on a topic of the experimenter's choosing. One of four speech topics will be conducted (counterbalanced). The investigators will measure participants' expectation that they will be negatively socially evaluated by the audience during the public speech. The investigators will measure this in anticipation of the speech (likelihood that the participant will be negatively socially evaluated) and after completing the speech (likelihood that the participant was negatively socially evaluated). Likelihood expectancy will be measured on a 0-100 scale, where 0 = certain they will not negatively evaluate you, 50 = completely uncertain, and 100 = certain they will negatively evaluate you. Higher = worse.
Behavioral Approach Task - Severity Expectancy | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Self-reported belief that, if participant will be / was negatively socially evaluated during public speaking Behavioral Approach Task, how severe do they think the negative social evaluation will be / was. The Behavioral Approach Task is a task in which the participant gives a speech to a small audience (1-4 people) on a topic of the experimenter's choosing. One of four speech topics will be conducted (counterbalanced). The investigators will measure participants' expectation that, if they are negatively socially evaluated by the audience during the public speech, how severe do they believe that severity will be / was. The investigators will measure this in anticipation of the speech (severity of negative social evaluation if it were to occur) and after completing the speech (severity of negative social evaluation if it did occur). Severity expectancy will be measured on a 0-100 scale, where 0 = not at all, 50 = moderate, and 100 = extreme. Higher = worse.
Behavioral Approach Task - Like/Dislike of Speech | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Self-reported liking/disliking of public speech. The Behavioral Approach Task is a task in which the participant gives a speech to a small audience (1-4 people) on a topic of the experimenter's choosing. One of four speech topics will be conducted (counterbalanced). After completing the speech, participants will rate how much they liked or disliked giving their public speech (-10 = dislike very much, 0 = neutral, +10 = like very much). Higher = better.
Behavioral Approach Task - Skin Conductance | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Skin conductance during Behavioral Approach Task. The Behavioral Approach Task is a task in which the participant gives a speech to a small audience (1-4 people) on a topic of the experimenter's choosing. One of four speech topics will be conducted (counterbalanced). Skin conductance is a physiological measure that will be analyzed during the speech anticipation period, where participants sit quietly for 2 minutes prior to giving their speech. The investigators will assess mean skin conductance level during this anticipation period minus their mean skin conductance level during a 2-minute baseline period prior to the speech task. Higher = worse.
Behavioral Approach Task - Electrocardiography HF-HRV | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Electrocardiography during Behavioral Approach Task. The Behavioral Approach Task is a task in which the participant gives a speech to a small audience (1-4 people) on a topic of the experimenter's choosing. One of four speech topics will be conducted (counterbalanced). Electrocardiography is a physiological measure that will be analyzed during the speech anticipation period, where participants sit quietly for 2 minutes prior to giving their speech. Using electrocardiography, the investigators will analyze high frequency heart rate variability (HF-HRV) during this anticipation period. Higher = better.
Behavioral Approach Task - Electrocardiography RMSSD HRV | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Electrocardiography during Behavioral Approach Task. The Behavioral Approach Task is a task in which the participant gives a speech to a small audience (1-4 people) on a topic of the experimenter's choosing. One of four speech topics will be conducted (counterbalanced). Electrocardiography is a physiological measure that will be analyzed during the speech anticipation period, where participants sit quietly for 2 minutes prior to giving their speech. Using electrocardiography, the investigators will analyze root mean square of successive differences (RMSSD) heart rate variability (HRV) during this anticipation period. Higher = better.
Behavioral Approach Task - Electrocardiography LF/HF-HRV | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Electrocardiography during Behavioral Approach Task. The Behavioral Approach Task is a task in which the participant gives a speech to a small audience (1-4 people) on a topic of the experimenter's choosing. One of four speech topics will be conducted (counterbalanced). Electrocardiography is a physiological measure that will be analyzed during the speech anticipation period, where participants sit quietly for 2 minutes prior to giving their speech. Using electrocardiography, the investigators will analyze low frequency divided by high frequency heart rate variability (LF/HF-HRV) during this anticipation period. Higher = worse.
Behavioral Approach Task - Speech Duration | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  How long the participant delivers their speech (between 0 and 5 minutes). The Behavioral Approach Task is a task in which the participant gives a speech to a small audience (1-4 people) on a topic of the experimenter's choosing. One of four speech topics will be conducted (counterbalanced). Participants can stop their speech whenever they choose to do so (e.g., if feeling anxious). Speech duration is a behavioral measure. Higher = better.

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Self-report measure of social anxiety. This measure is a 48-item questionnaire in which participants respond to how much fear or anxiety (0-3 scale, where = 0 none, 1 = mild, 2 = moderate, and 3 = severe) and how much they avoid (0-3, where 0 = never (0%), 1 = occasionally (1-33%), 2 = often (33-67%), and 3 = usually (67-100%) 24 social situations. Scores range 0-144. Higher = worse.
Dimensional Anhedonia Rating Scale (DARS) | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Self-report measure of anhedonia / reward processing. This is a questionnaire consisting of 17 items on a 0-4 scale (0 = not at all, 2 = moderately, 4 = very much) asking participants to name several positive activities and then to what degree they would have positive thoughts or emotions regarding those activities (e.g., how much they want to do those activities). Scores range 0-68. Higher = better.
Depression, Anxiety, and Stress Scale (DASS-21) | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24). Also Sessions 2, 4, 6, 8 of each therapy (corresponding to ~weeks 1, 2, 3, 4, 7, 8, 9, 10).
  Self-report measures of depression, anxiety, and stress. Scale consists of 21 items (7 depression, 7 anxiety, and 7 stress) rated on a 0-3 scale (0 = did not apply to me at all, 1 = applied to me at some degree or some of the time, 2 = applied to me to a considerable degree or a good part of time, and 3 = applied to me very much or most of the time). Total scores range 0-63; depression, anxiety, and stress subscale scores range 0-21 each. Higher = worse.
Positive Valence Systems Scale (PVSS) | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24). Also Sessions 2, 4, 6, 8 of each therapy (corresponding to ~weeks 1, 2, 3, 4, 7, 8, 9, 10).
  Self-report measure of anhedonia / reward processing. This is a questionnaire consisting of 21 items on a 1-9 scale (1 = extremely untrue of me, 5 = neutral, 9 = extremely true of me) with statements related to NIMH's positive valence systems (e.g., anticipation of reward, response to reward attainment). Mean scores range 1-9. Higher = better.
Positive and Negative Affect Schedule (PANAS) | Pre Tx (week 0), Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6), Post Tx-2 (after Exposure Therapy) (~week 12), 3-Month Follow-Up (~week 24).
  Self-report measure of positive and negative affect. This is a questionnaire consisting of 20 items on a 1-5 scale (1 = very slightly or not at all, 3 = moderately, 5 = extremely). Each item is a positive or negative emotion, and participants rate how much they experienced that emotion. Two subscales are scored: positive affect and negative affect. Each subscale's score ranges 10-50. For the positive affect subscale, higher = better. For the negative affect subscale, higher = worse.
Fear Conditioning - fMRI BOLD during shock omission | Pre Tx (week 0) and Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6).
  Neural responses (i.e., BOLD) measurement during shock omission in extinction phase. BOLD responses during this stimulus will be contrasted to BOLD responses during inter-trial intervals (ITIs), with a focus on reward neurocircuitry (e.g., striatum). For BOLD values in the reward circuitry, higher = better.
Fear Conditioning - fMRI BOLD during conditional stimuli | Pre Tx (week 0) and Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6).
  Neural responses (i.e., BOLD) measurement during acquisition and extinction phases to each conditional stimulus. BOLD responses during these stimuli will be contrasted to BOLD responses during inter-trial intervals (ITIs), with a focus on neurocircuitry involved in threat processing (e.g., amygdala) and inhibition (e.g., ventromedial prefrontal cortex). For BOLD values in the threat circuitry, higher = worse. For BOLD values in the inhibitory circuitry, higher = better.
Exposure Therapy - Perceived Historical Likelihood of Feared Outcome | Sessions 1-8 of Exposure Therapy (corresponding to ~weeks 7-10).
  Self-report questionnaire item asking participants across all of the public speeches they have ever given, how often does it feel like their feared outcome (e.g., social rejection) has occurred. Scale ranges 0-100 (0 = 0% of the time, 100 = 100% of the time). Higher = worse.
Exposure Therapy - Perceived Historical Severity of Feared Outcome | Sessions 1-8 of Exposure Therapy (corresponding to ~weeks 7-10).
  Self-report questionnaire item asking participants across all of the public speeches they have ever given, when their feared outcome has occurred (e.g., social rejection) how severe does it feel like it has been. Scale ranges 0-100 (0 = not at all, 50 = moderate, 100 = extreme). Higher = worse.
Exposure Therapy - Public Speaking Valence | Sessions 1-8 of Exposure Therapy (corresponding to ~weeks 7-10).
  Self-report questionnaire item asking participants how much they like or dislike giving public speeches. Scale ranges -10 to +10 (-10 = dislike very much, 0 = neutral, +10 = like very much). Higher = better.
Exposure Therapy - Exposure Likelihood Expectancy | Sessions 1-8 of Exposure Therapy (corresponding to ~weeks 7-10).
  Self-report questionnaire item asking participants how certain they are that their feared outcome will/did occur during a given exposure ranging 0-100 (0 = certain will/did not occur, 50 = completely uncertain, 100 = certain will/did occur). Higher = worse.
Exposure Therapy - Exposure Severity Expectancy | Sessions 1-8 of Exposure Therapy (corresponding to ~weeks 7-10).
  Self-report questionnaire item asking participants how severe they believe their feared outcome will be / was if it were to / did occur, ranging 0-100 (0 = not at all, 50 = moderate, 100 = extreme). Higher = worse.
Exposure Therapy - Exposure Fear/Anxiety | Sessions 1-8 of Exposure Therapy (corresponding to ~weeks 7-10).
  Self-report questionnaire item asking participants how their fear/anxiety level regarding a given exposure (0 = none, 50 = moderate, 100 = extreme). Higher = worse.
Exposure Therapy - Exposure Relief-Pleasantness | Sessions 1-8 of Exposure Therapy (corresponding to ~weeks 7-10).
  Self-report questionnaire item asking participants how relieved/pleasant they feel because their feared outcome (e.g., social rejection) did not occur or likely did not occur, ranging 0-100 (0 = not at all, 50 = moderately, 100 = extremely). Higher = better.
Exposure Therapy - Mood | Sessions 1-8 of Exposure Therapy (corresponding to ~weeks 7-10).
  Self-report questionnaire item asking participants their current mood, ranging -10 to +10 (-10 = extremely negative, = 0 neutral, +10 = extremely positive). Higher = better.
Positive Affect Treatment - Behavioral and Relaxation Treatment: Mood | Sessions 1-8 of Positive Affect Treatment - Behavioral or Relaxation Treatment (corresponding to ~weeks 1-4).
  Self-report questionnaire item asking participants their current mood, ranging -10 to +10 (-10 = extremely negative, = 0 neutral, +10 = extremely positive). Higher = better.
Exposure Therapy - EMA Likelihood Expectancy | Questionnaires are sent after each exposure therapy session: 2 hours after session, 24 hours after, and 48 hours after.
  Questionnaire item measured with regards to most recently completed exposure via ecological momentary assessment (EMA). Participant rates how certain they are that, if participant were to repeat the most recent exposure from their previous Exposure Therapy session, how certain are they that their feared outcome (e.g., social rejection) would occur. Scores range 0-100 (0 = certain will not occur, 50 = completely uncertain, 100 = certain will occur). Higher = worse.
Exposure Therapy - EMA Severity Expectancy | Questionnaires are sent after each exposure therapy session: 2 hours after session, 24 hours after, and 48 hours after.
  Questionnaire item measured with regards to most recently completed exposure via ecological momentary assessment (EMA). Participant rates, if they were to repeat the most recent exposure from their previous Exposure Therapy session and their feared outcome (e.g., social rejection) were to occur, how severe do they believe their feared outcome would be. Scores range 0-100 (0 = not at all, 50 = moderate, 100 = extreme). Higher = worse.
Exposure Therapy - EMA Fear/Anxiety | Questionnaires are sent after each exposure therapy session: 2 hours after session, 24 hours after, and 48 hours after.
  Questionnaire item measured with regards to most recently completed exposure via ecological momentary assessment (EMA). Participant rates, if they were to repeat the most recent exposure from their previous Exposure Therapy session, how much fear/anxiety would they have. Scores range 0-100 (0 = none, 50 = moderate, 100 = extreme). Higher = worse.
Exposure Therapy - EMA Relief-Pleasantness | Questionnaires are sent after each exposure therapy session: 2 hours after session, 24 hours after, and 48 hours after.
  Questionnaire item measured with regards to most recently completed exposure via ecological momentary assessment (EMA). Participant rates, if they were to repeat the most recent exposure from their previous Exposure Therapy session and their feared outcome (e.g., social rejection) were to not occur, how pleasant/relieved would they feel. Scores range 0-100 (0 = not at all, 50 = moderate, 100 = extreme). Higher = better.
Exposure Therapy - EMA Valence | Questionnaires are sent after each exposure therapy session: 2 hours after session, 24 hours after, and 48 hours after.
  Questionnaire item asking how much participant likes or dislikes giving public speeches. Scores range -10 to +10 (-10 = dislike very much, 0 = neutral, +10 = like very much). Higher = better.
Fear Conditioning - Likelihood Expectancy | Pre Tx (week 0) and Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6).
  During fear conditioning task, questionnaire item asking how certain the participant is that they will receive electric shock the next time they see each stimulus. Scores range 1-9 (1 = certain "no", 5 = completely uncertain, 9 = certain "yes"). Higher = worse.
Fear Conditioning - Severity Expectancy | Pre Tx (week 0) and Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6).
  During fear conditioning task, questionnaire item asking how certain the participant is that the next time they see each stimulus, if they were to receive electric shock, how severe do they believe it will be. Scores range 1-9 (1 = not at all, 5 = moderate, 9 = extreme). Higher = worse.
Fear Conditioning - Fear | Pre Tx (week 0) and Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6).
  During fear conditioning task, questionnaire item measured asking how fearful each stimulus makes them feel. Scores range 1-9 (1 = not at all, 5 = moderately, 9 = extremely). Higher = worse.
Fear Conditioning - Relief-Pleasantness | Pre Tx (week 0) and Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6).
  During fear conditioning task in the extinction phase, questionnaire item measuring how pleasant/relieved the participant feels because this stimulus did not result in electric shock. Scores range 1-9 (1 = not at all, 5 = moderately, 9 = very). Higher = better.
Fear Conditioning - Skin Conductance | Pre Tx (week 0) and Post Tx-1 (after PAT-B or Relaxation Treatment) (~week 6).
  During fear conditioning task, measure skin conductance (physiological) and calculate skin conductance response to each stimulus by subtracting the mean value 2sec prior to each stimulus from the maximum value 1-6sec after each stimulus's onset. Then, range correct the scores by dividing by the largest observed skin conductance value, and then normalizing the range-corrected scores by taking their square root. Scores range 0-1. Higher = worse.

CONTACTS AND LOCATIONS:
Overall Officials: Tomislav D Zbozinek, PhD, Principal Investigator — University of California, Los Angeles; Michelle G Craske, PhD, Study Chair — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to upload non-identifiable data to the National Institute of Mental Health's (NIMH) Data Archive (NDA) per their policy. This will include individual participant data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available on NDA per their requirements, starting January, 2025, and will remain there per NDA policy. Supporting Information will be available approximately around the time of completion of the clinical trial and be made available indefinitely.
Access Criteria: Access will be granted per NDA policy.

REFERENCES:
- See also: NIMH K23 grant — https://reporter.nih.gov/search/HYd0mkk89E6BrUefmDmi7A/project-details/10887339